CLINICAL TRIAL: NCT06274073
Title: Double-dorsal Versus Single-volar Digital Subcutaneous Anaesthetic Injection for Finger Injuries in the Emergency Department: A Randomised Controlled Trial
Brief Title: Double-dorsal Versus Single-volar Digital Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2-22-2566
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Laceration of Skin; Anesthesia, Local; Pain; Nerve Block
Keywords: Digital nerve block; Finger lacerations; Single palmar injection; Double dorsal injection; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Two parallel groups (two digital block techniques)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single injection palmar digital block (Experimental): The needle was inserted into the subcutaneous region from the palmar side to the root of the proximal phalanx, perpendicular to the frontal plane and the finger. For anesthesia, 3 ml of anesthetic agent (prilocaine hydrochloride) was applied to the described point with this single injection and the needle was slowly removed.
  Interventions: Procedure: Palmar digital block
- Double injection dorsal digital block (Experimental): The needle was inserted into the proximal dorsal root of the proximal phalanx, into both the medial and lateral parts, perpendicular to the fingers and the frontal plane. After the aspiration, the injection was performed slowly and the needle was withdrawn concurently. A total of 3 ml of anesthetic agent (prilocaine hydrochloride) was injected into both the medial and lateral parts of the finger, 1.5 ml for each side.
  Interventions: Procedure: Dorsal digital block

INTERVENTIONS:
Procedure: Dorsal digital block — Dorsal regional digital block anesthesia (No drug or device is being investigated here; the two digital block procedure mentioned are compared)
  Arms: Double injection dorsal digital block
Procedure: Palmar digital block — Palmar regional digital block anesthesia (No drug or device is being investigated here; the two digital block procedures mentioned are compared)
  Arms: Single injection palmar digital block

SUMMARY:
The aim of this study is to compare the traditional dorsal double injection digital block with the palmar single injection technique in the suturing of acute traumatic hand finger lacerations in terms of injection pain score (NRS), anesthesia onset time, and success of anesthesia.

It is understood that single injection digital block and double injection digital block techniques do not have significant advantages over each other in terms of pain levels and procedure times.

However, the need for rescue anesthesia was evaluated to be lower in the single injection digital block technique. This difference is especially due to measurements in the volar region incisions.

According to the results of this study, we think that choosing the single injection digital block technique for volar region incisions is a more rational approach, especially in terms of the data of the need for rescue anesthesia.

DETAILED DESCRIPTION:
Randomized, parallel controlled, open labeled experimental study

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years of age
* Isolated traumatic acute hand finger lacerations requiring suturing
* Admissions within 6 hours of injury
* Patients who can cooperate with the NRS score
* Patients who gave consent

Exclusion Criteria:

* Vein, nerve and tendon lacerations on the hand that require repair
* Amputation or bone fracture
* Those who have used analgesics in the last 12 hours
* Hemodynamically unstable patients
* Known allergy to prilocaine hydrochloride

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Anesthesia pain score | 3rd minute
  Numerical rating scale (NRS): 0 to 10 (min-max); higher scores indicates more pain

SECONDARY OUTCOMES:
Anesthesia onset time | Measurements are provided per 30 seconds (30-60-90-120 seconds and more if necessary)
  Time achieved to total anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Alp Şener, Assoc prof, Principal Investigator — Ankara Yıldırım Beyazıt University Faculty of Medicine
Locations (1):
- Ankara City Hospital Emergency Medicine Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No